CLINICAL TRIAL: NCT06990230
Title: Prospective, Multicenter, Randomized Controlled, Non-inferior Clinical Study to Evaluate the Safety and Efficacy of Radiofrequency Transseptal Puncture System in Atrial Septul
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Yibo Yu, Associate chief physician, First Affiliated Hospital of Ningbo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF20240131; FAHNBU20240581 (Other Grant/Funding Number: Heayoung Medical Technology (Suzhou) Co., Ltd)
Record Dates: First submitted 2025-03-10; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Evaluation of the Radiofrequency Transseptal Puncture System; Atrial Septum Puncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): RF Cross
  Interventions: Device: Radiofrequency Transseptal Puncture System and Auxiliary Device
- Control Group (Active Comparator): Braidin Cross
  Interventions: Device: Radiofrequency Transseptal Puncture System and Auxiliary Device

INTERVENTIONS:
Device: Radiofrequency Transseptal Puncture System and Auxiliary Device — The intervention in this study stands out due to its specific focus on evaluating the safety and efficacy of a radiofrequency transseptal puncture system designed exclusively for use in the atrial septum, with the purpose of establishing a passage from the right atrium to the left atrium. This system incorporates an auxiliary radiofrequency puncture device, which serves as a crucial supportive component, enhancing the overall functionality and precision of the primary transseptal puncture system.
  What further distinguishes this intervention from others is its utilization of radiofrequency energy to facilitate the transseptal puncture. Unlike traditional mechanical puncture methods, which can have a steep learning curve, potentially cause serious complications such as pericardial tamponade and cardiac rupture, and may be time-consuming and imprecise in predicting the puncture site, the radiofrequency puncture device provides a more controlled and predictable approach. The radiofrequenc

SUMMARY:
To evaluate the safety and efficacy of radiofrequency transseptal puncture system and its auxiliary radiofrequency puncture device in atrial septum.

Evaluation indicators:

Success rate of atrial septum; The time required to successfully complete the atrial septum; Rate of failed atrial septal puncture crossing to the contralateral group; Performance evaluation of an RF transseptal puncture system; The incidence of complications related to atrial septal puncture; Rates of adverse events; Rates of serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

Participants scheduled to undergo transseptal access interventional cardiology procedure; The subjects were informed of the nature of the study, understood the purpose of the clinical trial, voluntarily participated and signed an informed consent form.

Exclusion Criteria:

1. The presence of an intracardiac mass, thrombus or vegetation on echocardiography; Left atrial myxoma;
2. subjects with ASD occluder or patch implantation;
3. hemorrhagic or coagulopathy; Or there is contraindication to antithrombotic drugs;
4. acute myocardial infarction within 4 weeks;
5. end-stage heart failure (ACC/AHAD stage); Or after heart transplantation; Or waiting for a heart transplant;
6. history of cerebrovascular accident within 30 days;
7. pregnant and lactating women;
8. acute systemic infection or sepsis;
9. patients who have participated in any drug and/or medical device clinical trial within 1 month before this trial;
10. atrial septal puncture within 3 months;
11. life expectancy less than one year;
12. The investigator judged that the patient had poor compliance and could not complete the study according to the requirements; Or other circumstances in which the researcher considers the subject to be unsuitable for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Success rate of atrial septum | It is expected to last 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heayoung Medical Technology (Suzhou) Co., Ltd, Suzhou, Jiangsu, China